CLINICAL TRIAL: NCT04613141
Title: A Phase II Randomised Controlled Trial Comparing Home-based Self-managed Rehabilitation Program Using eHealth Technologies (Called WalkingTall-PD) With a Low-intensity Exercise Program (Called Mobility-plus).
Brief Title: The WalkingTall Study: Comparing WalkingTall With Parkinson's Disease (WalkingTall-PD) With Mobility-plus to Reduce Falls and Improve Mobility.
Acronym: WalkingTall-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Shake it up Australia Foundation (Unknown); Sensoria Health Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WalkingTallPD2019
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Falls; Step-time variability; Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessments that occur after baseline randomization will be completed by blinded assessor. Excluding the immediate effect of stimulation on step time variability, which is impossible to blind as the participant using a stimulation device, which is not practical to conceal.
  Statistician blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobility-plus (Sham Comparator): Mobility-plus is a "pseudo placebo" comparator program using non-slip socks, a low intensity paper-based exercise program and health information specific to Parkinson's Disease.
  Interventions: Other: Mobility-plus
- WalkingTall-PD (Experimental): WalkingTall-PD is a novel neuro-rehabilitation program delivered through a tablet/smart phone and smart garments (socks, insoles or ankle bands) for people with Parkinson's disease that aims to improve mobility and reduce falls. WalkingTall-PD combines a variety of PD-specific rhythmic stimuli (auditory, visual and haptic cues) which are synchronised with high intensity stepping, walking and balance training.
  Interventions: Device: WalkingTall-PD

INTERVENTIONS:
Device: WalkingTall-PD — Smart garment (socks, insoles or ankle bands) delivering rhythmic haptic stimuli to the ankle timed with preferred cadence. Smart phone application delivers auditory cues synchronised with haptic stimuli. Smart phone application delivers a neurorehabilitation program.
  Arms: WalkingTall-PD
Other: Mobility-plus — Active 'pseudo placebo' comparator using a paper-based body weight exercise program.
  Arms: Mobility-plus

SUMMARY:
The purpose of this study is to determine and compare the effectiveness of WalkingTall-PD (the new intervention) against Mobility-plus (a PD appropriate exercise program) with respect to stabilizing gait, reducing step-time variability, preventing falls and enhancing independence in people with Parkinson's disease.

WalkingTall-PD is a novel neuro-rehabilitation program delivered through a tablet/smart phone and smart socks for people with Parkinson's disease that aims to improve mobility and reduce falls. WalkingTall-PD combines a variety of PD-specific rhythmic stimuli (auditory, visual and haptic cues) which are synchronised with high intensity stepping, walking and balance training.

Mobility-plus is a "pseudo placebo" comparator program using non-slip socks, a low intensity paper-based exercise program and health information specific to Parkinson's Disease.

DETAILED DESCRIPTION:
WalkingTall-PD is designed to rehabilitate gait and balance in a minimum of 6-weeks (program progression and total duration is based on sessions completed). It uses affordable eHealth technologies (tablet, phone, smart socks or leg bands, depending on participant preference, with vibration motors, step mat and earbuds). Specific to Parkinson's disease (PD), it uses rhythmic cues to address excessive step-time variability, balance impairments and freezing of gait (FOG) (Henderson et al., 2017; Allen et al., 2013). The key aspect of this intervention is the stimulation provided by the smart socks/leg bands that vibrate. The stimulus duty cycle is synchronised with the participants walking gait to entrain neuromuscular signals and enhance sensorimotor integration. This results in an immediate improvement in motor control during gait, reduced movement variability and increased walking ability. The integration of our eHealth tools with home visits and telehealth appointments into a continuous user experience is another major strength of our program. Each component is introduced during 1:1 home visits and/or telehealth appointments to ensure standardization of the clinical trial and maximize the safety of participants. The home visits and/or telehealth appointments will be conducted by a trainer (physiotherapist or exercise physiologist with experience in working with people with PD).

WalkingTall-PD meets the urgent need for an effective, affordable and scalable self-managed eHealth solution for people with PD. It includes an evidence-based program to enhance independence and prevent falls. The scientific rationale and eHealth technology underpinning WalkingTall-PD are well tested. Our team has demonstrated that home-based approaches have high acceptability and adherence rates, shown that balance training can reduce fall-risk and that external cues can reduce step-time variability in people with PD. Participants may use their preferred devices (or devices we supply) to access WalkingTall-PD, which will be available across platforms. Components are introduced during 1:1 home visits and telehealth appointments by a trainer. Delivery is then unsupervised using self-management principles, with ongoing remote monitoring a web-based central monitoring platform and database back-end.Participants will be informed that WalkingTall-PD is a supplementary program and does not replace usual care. The WalkingTall-PD program comprises the following components:

(i) Balance training is introduced in the week-one home visit or telehealth appointment by the trainer using the WalkingTall smart phone app. Baseline balance ability is determined by completing a series of balance exercises using the app with supervision from the trainer. For participants who choose the telehealth option, the primary device (smart phone) will provide the training program while a secondary device (iPad) will be used for patient safety monitoring and telehealth consultation. Exercises include heel raises, postural transitions, reaching and stepping in different directions and holding poses that challenge balance. Props used include a mobile stand (primary device), a tablet stand for the secondary device, non-slip balance mat and chairs for support. Balance training starts with simple movement sequences and progresses to more challenging balance poses based on participant feedback. Movements during balance training are guided by the combination of haptic cues provided by the smart socks, insoles or ankle bands(with the choice of smart garment based on participant preference), auditory cues by the phone app and visual cues by the balance/stepping mat. Participants will be encouraged to complete 5 by 10-minutes balance training sessions/week. Participants who choose the telehealth option will be provided with a home visit if they have difficulty with the balance training.

(ii) Walk training (in a safe environment) is introduced in the second home visit or telehealth appointment (no sooner than week-3) by the trainer using our WalkingTall phone app. Participant-adjustable rhythmic cues (Brodie et al., 2015) auditory, visual and haptic cues are used to reduce gait variability during gait training. Participants are instructed how to select an appropriate walking course (clear of trip hazards and with appropriate rest areas), target cadence and training/rest duration by the trainer. The walking course will be approved by the trainers, either in person or remotely via video recording if the participant chooses the telehealth option. For participants included in the telehealth option, if the trainer has concerns about the selected walking track, a home visit will be provided to fix any safety issues. Each session, consists of 5 by 2-minutes walks with 30-seconds rest between each walk. Rhythmic auditory cues (self-selected metronome) are provided by the phone app and earbuds can be used for discretion. Rhythmic haptic cues are provided by the smart socks, insoles or smart ankle bands, with the choice of smart garment based on participant preference. Participant-specific visual cues may also be used, if required, such as parallel lines fixed perpendicular to the walking track to step over. Participants will be instructed to use their normal walking aids as appropriate. Participants will be encouraged to complete 5 by 10-minute walk training in addition to the 5 by 10-minute balance training sessions each week. Participants who choose the telehealth option will be provided with a home visit if they have difficulty with the walk training.

(iii) Step training is introduced in the third home visit or telehealth appointment (no sooner than week-5) by the trainer using the WalkingTall phone app. Visual, auditory and haptic cues are synchronized with the movement to retrain impaired stepping (Caetano et al., 2018), turning, balance (Allen et al., 2013) and strength in people with PD. Auditory stepping cues are provided by the phone app using a metronome beat. Visual cues are provided by the non-slip stepping mat. Haptic stepping cues are provided by small vibrators. Participants will be encouraged to complete 5 by 10-minute step/strength training, 5 by 10-minute walk training and 5 by 10-minute balance training sessions each week. In week-5 the trainer will also introduce walk training in more complex environments or walking as part of normal daily-life activities as appropriate. Participants who choose the telehealth option will be provided with a home visit if they have difficulty with the step and training.

(iv) Post intervention. Reassessment will occur at 3-months. (v) Continuity of care is is provided by WalkingTall-PD using the WalkingTall phone app to self-manage any ongoing gait and balance impairments. Following the reassessment, participants will receive another home visit or telehealth consultation where an individualised program will be prescribed based on participant preference. For the remainder of the 3-months, participants will then be encouraged to complete at least 3 sessions per week of their individually prescribed WalkingTall-PD program. Training targets will be set and reviewed via monthly teleconferences and using the WalkingTall Study "Monthly Progress Chart". A study hotline is provided.

Mobility-plus is a "pseudo placebo" comparator program. It is not a true placebo because participants will be aware of which program they are in. However, both programs comprise of components that have potential to improve mobility and reduce falls risk and participants will not be informed of our hypothesis that WalkingTall-PD will be more effective than Mobility-plus. Participants in the Mobility-plus group will also be provided with gait-specific exercise equipment (two pairs of non-slips socks, which provide increased foot sensation through a pattern of raise non-slip nodules), a low intensity exercise program (3sessions per week) and health information specific to PD (included in the training manual). Participants will be informed that Mobility-plus is a supplementary program and does not replace usual care. The Mobility-plus program comprises the following components:

(i) Mobility exercises are introduced in week-1 by the trainer using the Mobility-plus exercise manual.Mobility-plus participants are provided with two pairs of non-slips socks and instructed to wear them while completing the Mobility-plus exercises. Participants use a chair as a prop and for balance support. Exercises include: (1) Standing hip abduction; (2) Standing knee flexion; (3) Seated knee extension; (4) Standing hip extension; and, (5) Standing hip flexion. Participants are instructed to complete 3-sets of 10-reps, for each exercise, for each leg, 3 times per week. Each session lasts approximately 10-minutes. For participants who choose the telehealth option this will be done via video conferencing and participants will be provided with a home visit if they have difficulty with the exercises.

(ii) Post intervention. Reassessment will occur at 3-months. (iii) Continuity of care is provided through the Mobility-plus manual. Participants will be encouraged to keep doing their Mobility-plus exercises 3 times per week for the remainder of the 3-month program. A study hotline is also provided for the Mobility-plus group.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with idiopathic Parkinson's disease (according to UK PD Society Brain Bank Criteria);
* Mild to severe (Hoehn and Yahr stage 1-4 idiopathic Parkinson's disease;
* Ability to walk 18 meters with or without an aid;
* At least one fall in the past 6 months, or at least 2 falls in the past 12 months, or severe mobility impairment such as freezing of gait, or history of near falls.
* Being stable on anti-Parkinsonian medications for > 1 month;
* Living independently in the community or retirement village;
* Able to communicate in English language.

Exclusion Criteria:

* Diagnosis of other neurological and/ or significant cognitive impairments (Montreal Cognitive Assessment < 19 points);
* Atypical Parkinsonism;
* Less than 6 months post deep brain stimulation surgery;
* Excessively high fall rates (> 12 falls in the past 6 months);
* Insufficient foot/ ankle sensation;
* Do not speak English;
* Have another medical condition besides Parkinson's disease that significantly impairs mobility, balance or ability to exercise safely;
* Already participating in a different study to improve mobility or prevent falls.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Gait variability (immediate effect of stimulation) | Baseline and 3-month re-assessment
  Standard deviation of step times will be assessed by a wearable device (McRoberts). This will be measured for both face-to-face and telehealth options. Baseline walking is compared to baseline walking with simulation (for the intervention group) and compared to walking with non-slip socks (for the control group). This will be repeated at 3-months. For face to face, gait variability will be assessed using the middle 16m of 4 x 20m straight line walks. For telehealth, it may not be possible to find a 20m straight line walking track, in which case more laps will be required to get a total distance of at least 80 meters. Regardless of the face to face or telehealth option, the same walking track will be used by each participant for each assessment to ensure consistency.
Gait variability (no stimulation) | Baseline and 3-month re-assessment
  Standard deviation of step times will be assessed by a wearable device (McRoberts). This will be measured for both face-to-face and telehealth options. For both baseline and re-assessment the no stimulation condition is used. For face to face, gait variability will be assessed using the middle 16m of 4 x 20m straight line walks. For telehealth, it may not be possible to find a 20m straight line walking track, in which case more laps will be required to get a total distance of at least 80 meters. Regardless of the face to face or telehealth option, the same walking track will be used by each participant for each assessment to ensure consistency.

SECONDARY OUTCOMES:
Rate of falling | Baseline and post-intervention (3-months)
  Rate of falling will be ascertained using weekly electronic falls calendars and email reminders. This will be measured for both face-to-face and telehealth options.
Levodopa equivalency daily dosage | Baseline and post-intervention (3-months)
  This will be measured for both face-to-face and telehealth options.
Postural balance and mobility | Baseline and post-intervention (3-months)
  Postural balance and mobility using the Mini-best test. This will be measured for both face-to-face and telehealth options. Although, this assessment will be adapted for telehealth purpose. Only items that are safer to be undertaken without a therapist support will be performed.
Physical activity enjoyment | Post-intervention (3-months)
  Physical activity enjoyment will be assessed using Physical Activity Enjoyment Scale Questionnaire. This will be measured for both face-to-face and telehealth options.
System usability | Post-intervention (3-months)
  System usability will be assessed using System Usability Scale Questionnaire. This will be measured for both face-to-face and telehealth options, and only for individuals who will receive the Walking-Tall PD training.
Attitudes to fall related intervention | Post-intervention (3-months)
  Attitudes to fall related intervention will be assessed using Attitudes to Fall Related Intervention Scale Questionnaire. This will be measured for both face-to-face and telehealth options.
Exercise self-efficacy | Post-intervention (3-months)
  Exercise self-efficacy will be assessed using Exercise Self-Efficacy Scale Questionnaire. This will be measured for both face-to-face and telehealth options.
Health-related quality of life | Baseline and post-intervention (3-months)
  Health-related quality of life will be assessed using the European Quality of Life-5 EQ-5D. This will be measured for both face-to-face and telehealth options.
Parkinson's disease health status | Baseline and post-intervention (3-months)
  Parkinson's disease health status using a PD-specific quality-of-life questionnaire. This will be measured for both face-to-face and telehealth options.
Lower extremity physical performance | Baseline and post-intervention (3-months)
  Lower extremity physical performance will be assessed using the Short Physical Performance Battery. This will be measured for both face-to-face and telehealth options.
Parkinson's disease symptoms | Baseline and post-intervention (3-months)
  Parkinson's disease symptoms will be assessed using the Movement Disorders Society - Unified Parkinson's Disease Rating Scale. This will be measured for both face-to-face and telehealth options. Although, this assessment will be adapted for telehealth purpose.
Freezing of gait | Baseline and post-intervention (3-months)
  Freezing of gait will be assessed using the New Freezing of Gait Questionnaire. This will be measured for both face-to-face and telehealth options.
Concern about falling | Baseline and post-intervention (3-months)
  Concern about falling will be assessed using the Iconographical Falls Efficacy Scale Questionnaire. This will be measured for both face-to-face and telehealth options.
Physical activity level | Baseline and post-intervention (3-months)
  Activity levels will be assessed using the Incidental and Planned Exercise Questionnaire. This will be measured for both face-to-face and telehealth options.
Activity of daily living | Baseline and post-intervention (3-months)
  Activities of daily living will be assessed using 1-week remote monitoring, including total steps/day, step-time variability, uninterrupted walk durations, falls, near falls and freezing of gait events. This will be measured for both face-to-face and telehealth options.
Exercise adherence | Post-intervention (3-months)
  Exercise adherence will be assessed using monthly exercise calendars. An e-mail with a web link will be send to the participants, and they will be asked to report if any falls happened in a previous month. This will be measured for both face-to-face and telehealth options.
Health service use | Post-intervention (3-months)
  Health service use will be assessed using a monthly questionnaire. This will be measured for both face-to-face and telehealth options.
Freezing of gait | Baseline and post-intervention (3-months)
  Freezing of gait will be assessed by a wearable device during a freezing of gait elicitation protocol. This will be only measured for the face-to-face option.
Simple stepping ability | Baseline (week 1) and post-intervention (7 weeks after randomisation).
  Simple stepping ability and reaction time will be assessed using the choice stepping reaction time test.
  They will be only measured for face-to-face option.
Inhibitory stepping ability | Baseline and post-intervention (3-months)
  Inhibitory stepping ability and reaction time will be assessed using the inhibitory choice stepping reaction time test.
  They will be only measured for face-to-face option.
Complex stepping ability | Baseline and post-intervention (3-months)
  Complex stepping ability and reaction time will be assessed using the stroop stepping test.
  They will be only measured for face-to-face option.
Polypharmacy | Baseline and post-intervention (3-months)
  Change in polypharmacy (the amount of medication taken). This will be measured for both face-to-face and telehealth options.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Brodie, Dr, Principal Investigator — The University of New South Wales
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886